CLINICAL TRIAL: NCT01328626
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABT-199 in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia and Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M12-175
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Chronic Lymphocytic Leukemia; Non-Hodgkin Lymphoma
Keywords: Safety; Maximum Tolerated Dose; Pharmacokinetics; ABT-199; Preliminary Efficacy; Cancer; Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Neoplasms | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (CLL/SLL subjects) (Experimental): Chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL) subjects
  Interventions: Drug: ABT-199
- Arm B (NHL subjects) (Experimental): Non-Hodgkin lymphoma (NHL) subjects
  Interventions: Drug: ABT-199

INTERVENTIONS:
Drug: ABT-199 — Arm A (Cohorts 1-8) and Arm B (Cohort 1-6): Subjects in dose escalation phase will receive 1 dose of ABT-199, followed by 6 days off drug, followed by continuous once daily dosing with ABT-199. Arm B (Cohorts 7+): Subjects in dose escalation phase will receive continuous once daily dosing with ABT-199. Arm A and Arm B: Subjects in expanded safety cohort will receive continuous once daily dosing with ABT-199.

SUMMARY:
This is a Phase 1, open-label, multicenter study evaluating the safety and PK profile of ABT-199 under a once daily dosing schedule. Two arms will be implemented for dose escalation: Arm A, CLL/SLL subjects and Arm B, NHL subjects. Arm A is designed to enroll approximately 116 subjects with relapsed or refractory CLL or SLL and Arm B is designed to enroll approximately 95 subjects with relapsed or refractory NHL. Fifty-six subjects were enrolled in Arm A and approximately 55 subjects will be enrolled in Arm B during the dose escalation portion of the study, with the objective of defining dose limiting toxicities (DLTs) and the MTD. Once the MTD is declared for the arm, approximately 60 additional CLL/SLL subjects in Arm A and approximately 20 additional DLBCL subjects and 20 additional follicular lymphoma subjects in Arm B will be enrolled in an expanded safety portion of the study at the recommended phase 2 dose (RPTD) and schedule.

DETAILED DESCRIPTION:
Interventional Study Design - Primary Purpose: Determination of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have either:

  * (Arm A) relapsed or refractory CLL/SLL and require treatment in the opinion of the Investigator. Subject must have relapsed following or be refractory to standard treatments such as fludarabine based regimens (F, FC, FR, FCR) or alkylator (chlorambucil, bendamustine) based regimens. In addition, there are no other curative options, and the subject has exhausted options that would be considered standard of care, or
  * (Arm B) relapsed or refractory NHL and require treatment in the opinion of the Investigator. Subject must have histologically documented diagnosis of NHL as defined in the World Health Organization classification scheme, except as noted in the exclusion criteria. Subject must have relapsed following or be refractory to standard treatments such as R-CHOP, R-CVP, or fludarabine based regimens. In addition, there are no other curative options, and the subject has exhausted options that would be considered standard of care. Subjects with other lymphoproliferative diseases can be considered in consultation with the Abbott medical monitor.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance score less than or equal to 1.
* Subject must have adequate bone marrow independent of growth factor support per local laboratory reference range at Screening.
* Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening.

Exclusion Criteria:

* CLL subject has undergone an allogeneic or autologous stem cell transplant or NHL subject has undergone an allogeneic stem cell transplant or has been diagnosed with Post-Transplant Lymphoproliferative Disease, Burkitt's lymphoma, Burkitt-like lymphoma, or lymphoblastic lymphoma/leukemia.
* Subject has tested positive for HIV.
* Subject has a cardiovascular disability status of New York Heart Association Class greater or equal to 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity, results in fatigue, palpitations, dyspnea or anginal pain.
* Subject has a significant history of renal, neurologic, psychiatric, pulmonary, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the Investigator would adversely affect his/her participating in this study.
* Subject has received a monoclonal antibody for anti-neoplastic intent within 8 weeks prior to the first dose of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Determination of dose limiting toxicity (DLT), maximum tolerated dose (MTD), recommended phase two dose (RPTD), and lead-in period regimen | Lead-in period (2-5 weeks) plus 3 weeks of study drug administration at the designated cohort dose (continuous dosing)
  Protocol-defined events, which can not be attributed by the investigator to a clearly identifiable cause such as tumor progression, underlying illness, concurrent illness, or concomitant medication, will be considered a DLT. Dose limiting toxicities of tumor lysis syndrome observed during the lead-in period will be attributed to the lead-in period.
Number of subjects with adverse events | First 16 weeks of study drug administration and every 4 weeks thereafter (continuous dosing for an anticipated maximum duration of 9 months)
Determination of plasma peak concentration (Cmax) of ABT-199 | Up to Week 24 for ABT-199
  Blood and urine samples for pharmacokinetic analysis of ABT-199 will be collected at designated time points
Determination of trough concentration (Ctrough) of ABT-199 | Up to Week 24 for ABT-199
  Blood and urine samples for pharmacokinetic analysis of ABT-199 will be collected at designated time points
Determination of area under the concentration versus time curve (AUC) of ABT-199 | Up to Week 24 for ABT-199
  Blood and urine samples for pharmacokinetic analysis of ABT-199 will be collected at designated time points

SECONDARY OUTCOMES:
Food Effect - Cmax | Approximately 3 days
  Pharmacokinetic (PK) parameter Cmax (maximum plasma concentration of ABT-199) between each diet (ABT-199 under fasting versus low-fat, and fasting versus high-fat conditions (Cohorts 1-6 in Arm B subjects only)
Preliminary efficacy assessment | Starting Week 4 for clinical disease progression and Week 6 for tumor response; and every 4 weeks thereafter (continuous dosing for an anticipated maximum duration of 9 months)
  Tumor response or clinical disease progression
Minimal residual disease collection (MRD) | At least 2 months after the CR, CRi criteria for tumor response are first met. Every 12 weeks thereafter, until MRD negativity has been achieved (in peripheral blood).
  MRD assessed in the peripheral blood and/or bone marrow (BM) either by four color flow cytometry or ASO-PCR, will be measured in CLL subjects achieving CR/CRi.
Food Effect - Tmax | Approximately 3 days
  Pharmacokinetic (PK) parameter Tmax (time to reach maximum plasma concentration of ABT-199) between each diet (ABT-199 under fasting versus low-fat, and fasting versus high-fat conditions (Cohorts 1-6 in Arm B subjects only)
Food Effect - AUC | Approximately 3 days
  Pharmacokinetic (PK) parameter AUC (area under the concentration-time curve from time zero to hour 24 of ABT-199) between each diet (ABT-199 under fasting versus low-fat, and fasting versus high-fat conditions (Cohorts 1-6 in Arm B subjects only)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (10):
- United States (8):
  - University of Arizona Cancer Center - North Campus /ID# 52902, Tucson, Arizona
  - Ucsd /Id# 48325, La Jolla, California
  - Dana-Farber Cancer Institute /ID# 48324, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center /ID# 56810, New York, New York
  - University of Texas MD Anderson Cancer Center /ID# 48326, Houston, Texas
  - Swedish Medical Center /ID# 135853, Seattle, Washington
  - Fred Hutchinson Cancer Research /ID# 52882, Seattle, Washington
  - Univ of Wisconsin Hosp/Clinics /ID# 56811, Madison, Wisconsin
- Australia (2):
  - Peter MacCallum Cancer Ctr /ID# 48323, Melbourne, Victoria
  - Royal Melbourne Hospital /ID# 48322, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davids MS, Roberts AW, Seymour JF, Pagel JM, Kahl BS, Wierda WG, Puvvada S, Kipps TJ, Anderson MA, Salem AH, Dunbar M, Zhu M, Peale F, Ross JA, Gressick L, Desai M, Kim SY, Verdugo M, Humerickhouse RA, Gordon GB, Gerecitano JF. Phase I First-in-Human Study of Venetoclax in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma. J Clin Oncol. 2017 Mar 10;35(8):826-833. doi: 10.1200/JCO.2016.70.4320. Epub 2017 Jan 17. PMID 28095146
- [Derived] Davids MS, Roberts AW, Kenkre VP, Wierda WG, Kumar A, Kipps TJ, Boyer M, Salem AH, Pesko JC, Arzt JA, Mantas M, Kim SY, Seymour JF. Long-term Follow-up of Patients with Relapsed or Refractory Non-Hodgkin Lymphoma Treated with Venetoclax in a Phase I, First-in-Human Study. Clin Cancer Res. 2021 Sep 1;27(17):4690-4695. doi: 10.1158/1078-0432.CCR-20-4842. Epub 2021 Jun 3. PMID 34083230
- [Derived] Roberts AW, Ma S, Kipps TJ, Coutre SE, Davids MS, Eichhorst B, Hallek M, Byrd JC, Humphrey K, Zhou L, Chyla B, Nielsen J, Potluri J, Kim SY, Verdugo M, Stilgenbauer S, Wierda WG, Seymour JF. Efficacy of venetoclax in relapsed chronic lymphocytic leukemia is influenced by disease and response variables. Blood. 2019 Jul 11;134(2):111-122. doi: 10.1182/blood.2018882555. Epub 2019 Apr 25. PMID 31023700
- [Derived] Roberts AW, Davids MS, Pagel JM, Kahl BS, Puvvada SD, Gerecitano JF, Kipps TJ, Anderson MA, Brown JR, Gressick L, Wong S, Dunbar M, Zhu M, Desai MB, Cerri E, Heitner Enschede S, Humerickhouse RA, Wierda WG, Seymour JF. Targeting BCL2 with Venetoclax in Relapsed Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jan 28;374(4):311-22. doi: 10.1056/NEJMoa1513257. Epub 2015 Dec 6. PMID 26639348
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M12-175&Latitude=&Longitude=&LocationName=#additional-resources-section